CLINICAL TRIAL: NCT00572195
Title: RNS® System Long-term Treatment (LTT) Clinical Investigation
Brief Title: RNS® System LTT Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NeuroPace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP10005; P100026 (Other: United States FDA)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Responsive neurostimulation; RNS System; NeuroPace; Brain stimulation; Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Evaluation Group (stimulation ON) (Experimental): Group of subjects that have an RNS® System implanted, completed the RNS® System Pivotal or Feasibility study, and elected to continue to receive RNS® System responsive stimulation for the long term.
  Interventions: Device: RNS® System

INTERVENTIONS:
Device: RNS® System — The previously implanted RNS® System is programmed to provide responsive stimulation. Upon detecting electrographic patterns, previously identified by the neurologist or neurosurgeon as abnormal, the Neurostimulator provides brief pulses of electrical stimulation through the Leads to interrupt those patterns. Patients with epilepsy treated with responsive direct-brain stimulation with the RNS System typically receive less than 6 minutes of stimulation a day.

SUMMARY:
The RNS® System LTT study is designed to assess the ongoing safety and to evaluate the long-term efficacy of the RNS® System as an adjunctive therapy in reducing the frequency of seizures in individuals 18 years of age or older with partial onset seizures that are refractory to two or more antiepileptic medications. Candidates will continue to receive their epilepsy medications while participating in the trial.

DETAILED DESCRIPTION:
NeuroPace, Inc. is sponsoring an investigational device study of the RNS® System, the first closed loop responsive brain stimulator designed to treat refractory epilepsy. The RNS® System LTT study is an open-label multi-center prospective 7-year clinical investigation which follows completion of the RNS® System Pivotal or Feasibility study. Data regarding safety and efficacy are collected at 6-month intervals, and data regarding quality of life are collected at yearly intervals.

The study is designed to assess the ongoing safety and to evaluate the long-term efficacy of the RNS® System as an adjunctive therapy in reducing the frequency of medically uncontrolled and disabling partial onset seizures that start from one or two areas of the brain.

The RNS® System LTT study will provide additional data on the safety and efficacy of the RNS® System for 7 years following a subject's completion of the RNS® System Feasibility or Pivotal studies. Data from the RNS® System LTT study will be combined with data collected during the RNS® System Feasibility and Pivotal studies, resulting in 9 total years of post-implant follow-up data. These data will be used to calculate long-term SAE rate, percent change in seizure frequency (from pre-implant baseline), as well as the frequency of sudden unexplained death in epilepsy (SUDEP).

The RNS® Neurostimulator (a pacemaker-like device) and NeuroPace® Leads (tiny wires with electrodes) are implanted in the head. The Neurostimulator is a battery powered, microprocessor controlled device that detects and stores records of electrographic patterns (such as epileptiform, or seizure-like, activity) from the Leads within the brain. When the device detects an electrographic pattern, it responds by sending electrical stimulation through the Leads to a small part of the patient's brain to interrupt the electrographic pattern. This type of treatment is called responsive stimulation, but it is not yet known if it will work for the treatment of epilepsy. Direct brain stimulation therapy has already received approval in the United States, Europe, Canada, and Australia for the treatment of Essential Tremor and Parkinson's disease. Direct brain stimulation is not approved for the treatment of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has completed either the RNS® System Pivotal or Feasibility study
2. Subject has an implanted RNS® System
3. Subject has elected to continue to receive responsive neurostimulation therapy after completion of the RNS® System Pivotal or Feasibility study
4. Subject is able to attend scheduled appointments for the RNS® System LTT study

Exclusion Criteria:

1. Subject has active psychiatric or medical illness that makes it inadvisable for the subject to continue to receive responsive neurostimulation therapy with the RNS® System
2. Subject has been diagnosed with psychogenic or non-epileptic seizures, or primarily generalized seizures during the RNS® System Pivotal or Feasibility study
3. Subject has been noncompliant with scheduled appointments during the RNS® System Pivotal or Feasibility study
4. Subject has been noncompliant with maintaining seizure diaries during the RNS® System Pivotal or Feasibility study
5. Informed consent cannot be obtained from subject or caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2006-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha J Morrell, MD, Study Director — NeuroPace, Inc.
Locations (33):
- United States (33):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida at Gainesville, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia / Georgia Regents University, Augusta, Georgia
  - Rush University Medical Center / Epilepsy Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Via Christi Comprehensive Epilepsy Center, Wichita, Kansas
  - Louisiana State University Epilepsy Center of Excellence, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University / Columbia Presbyterian Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Background] Heck CN, King-Stephens D, Massey AD, Nair DR, Jobst BC, Barkley GL, Salanova V, Cole AJ, Smith MC, Gwinn RP, Skidmore C, Van Ness PC, Bergey GK, Park YD, Miller I, Geller E, Rutecki PA, Zimmerman R, Spencer DC, Goldman A, Edwards JC, Leiphart JW, Wharen RE, Fessler J, Fountain NB, Worrell GA, Gross RE, Eisenschenk S, Duckrow RB, Hirsch LJ, Bazil C, O'Donovan CA, Sun FT, Courtney TA, Seale CG, Morrell MJ. Two-year seizure reduction in adults with medically intractable partial onset epilepsy treated with responsive neurostimulation: final results of the RNS System Pivotal trial. Epilepsia. 2014 Mar;55(3):432-41. doi: 10.1111/epi.12534. Epub 2014 Feb 22. PMID 24621228
- [Background] Morrell MJ; RNS System in Epilepsy Study Group. Responsive cortical stimulation for the treatment of medically intractable partial epilepsy. Neurology. 2011 Sep 27;77(13):1295-304. doi: 10.1212/WNL.0b013e3182302056. Epub 2011 Sep 14. PMID 21917777
- [Result] Bergey GK, Morrell MJ, Mizrahi EM, Goldman A, King-Stephens D, Nair D, Srinivasan S, Jobst B, Gross RE, Shields DC, Barkley G, Salanova V, Olejniczak P, Cole A, Cash SS, Noe K, Wharen R, Worrell G, Murro AM, Edwards J, Duchowny M, Spencer D, Smith M, Geller E, Gwinn R, Skidmore C, Eisenschenk S, Berg M, Heck C, Van Ness P, Fountain N, Rutecki P, Massey A, O'Donovan C, Labar D, Duckrow RB, Hirsch LJ, Courtney T, Sun FT, Seale CG. Long-term treatment with responsive brain stimulation in adults with refractory partial seizures. Neurology. 2015 Feb 24;84(8):810-7. doi: 10.1212/WNL.0000000000001280. Epub 2015 Jan 23. PMID 25616485
- [Derived] Nair DR, Laxer KD, Weber PB, Murro AM, Park YD, Barkley GL, Smith BJ, Gwinn RP, Doherty MJ, Noe KH, Zimmerman RS, Bergey GK, Anderson WS, Heck C, Liu CY, Lee RW, Sadler T, Duckrow RB, Hirsch LJ, Wharen RE Jr, Tatum W, Srinivasan S, McKhann GM, Agostini MA, Alexopoulos AV, Jobst BC, Roberts DW, Salanova V, Witt TC, Cash SS, Cole AJ, Worrell GA, Lundstrom BN, Edwards JC, Halford JJ, Spencer DC, Ernst L, Skidmore CT, Sperling MR, Miller I, Geller EB, Berg MJ, Fessler AJ, Rutecki P, Goldman AM, Mizrahi EM, Gross RE, Shields DC, Schwartz TH, Labar DR, Fountain NB, Elias WJ, Olejniczak PW, Villemarette-Pittman NR, Eisenschenk S, Roper SN, Boggs JG, Courtney TA, Sun FT, Seale CG, Miller KL, Skarpaas TL, Morrell MJ; RNS System LTT Study. Nine-year prospective efficacy and safety of brain-responsive neurostimulation for focal epilepsy. Neurology. 2020 Sep 1;95(9):e1244-e1256. doi: 10.1212/WNL.0000000000010154. Epub 2020 Jul 20. PMID 32690786
- [Derived] DiLorenzo DJ, Mangubat EZ, Rossi MA, Byrne RW. Chronic unlimited recording electrocorticography-guided resective epilepsy surgery: technology-enabled enhanced fidelity in seizure focus localization with improved surgical efficacy. J Neurosurg. 2014 Jun;120(6):1402-14. doi: 10.3171/2014.1.JNS131592. Epub 2014 Mar 21. PMID 24655096

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evaluation Group (Stimulation ON)
Started | 230
Completed | 162
Not Completed | 68
Not completed — Withdrawal by Subject | 50
Not completed — Death | 9
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Evaluation Group (Stimulation ON)
Number analyzed (Participants) | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 223
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: The number of subjects having an SAE during the RNS® System LTT study.
Time Frame: 2 years post-implant through 9 years post-implant (7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation Group (Stimulation ON)
Number analyzed (Participants) | 230
Participants | 177
Statistical Analysis 1: Comparison: Evaluation Group (Stimulation ON); Test type: Other; Wilson score interval = 77, 95% CI 2-sided [71.1 to 81.9] — The value is for all serious adverse events, regardless of device relation; 95% confidence interval estimated using the Wilson score interval

2. Primary Outcome: Percentage Change From Baseline in Seizure Frequency
Description: The average percentage change in the mean frequency of total disabling seizures relative to pre-implant baseline. The percent change will be calculated for each subject over 6-month intervals beginning 6 months after RNS® System implant and continuing through completion of the RNS® System LTT study.
Time Frame: 6 months post-implant through 9 years post-implant (8.5 years)
Population: N represents the number of subjects who have data during that period.
Measure: Median (Inter-Quartile Range); unit: Percentage of Change
Arm/Group | Evaluation Group (Stimulation ON)
Number analyzed (Participants) | 230
Percentage of Change
  6-12 Months: number analyzed (Participants) | 229
  6-12 Months | -31.5 [-62.4 to -5.0]
  12-18 Months: number analyzed (Participants) | 229
  12-18 Months | -46.2 [-72.3 to -15.1]
  18-24 Months: number analyzed (Participants) | 229
  18-24 Months | -46.7 [-74.9 to -16.1]
  24-30 Months: number analyzed (Participants) | 223
  24-30 Months | -50.3 [-79.2 to -16.9]
  30-36 Months: number analyzed (Participants) | 218
  30-36 Months | -58.3 [-83.3 to -21.6]
  36-42 Months: number analyzed (Participants) | 218
  36-42 Months | -61.1 [-84.9 to -27.8]
  42-48 Months: number analyzed (Participants) | 209
  42-48 Months | -61.7 [-87.6 to -27.7]
  48-54 Months: number analyzed (Participants) | 201
  48-54 Months | -60.5 [-85.2 to -22.0]
  54-60 Months: number analyzed (Participants) | 198
  54-60 Months | -63.1 [-90.7 to -23.5]
  60-66 Months: number analyzed (Participants) | 190
  60-66 Months | -65.4 [-92.7 to -23.7]
  66-72 Months: number analyzed (Participants) | 185
  66-72 Months | -67.7 [-93.8 to -36.2]
  72-78 Months: number analyzed (Participants) | 181
  72-78 Months | -71.0 [-95.5 to -29.4]
  78-84 Months: number analyzed (Participants) | 178
  78-84 Months | -72.8 [-95.4 to -27.7]
  84-90 Months: number analyzed (Participants) | 171
  84-90 Months | -69.7 [-94.6 to -30.4]
  90-96 Months: number analyzed (Participants) | 171
  90-96 Months | -73.1 [-94.4 to -38.7]
  96-102 Months: number analyzed (Participants) | 168
  96-102 Months | -72.1 [-96.1 to -41.3]
  102-108 Months: number analyzed (Participants) | 158
  102-108 Months | -74.5 [-97.5 to -43.2]
  108-114 Months: number analyzed (Participants) | 110
  108-114 Months | -85.9 [-100.0 to -43.9]
  114-120 Months: number analyzed (Participants) | 30
  114-120 Months | -77.7 [-100.0 to -42.7]
  120-126 Months: number analyzed (Participants) | 12
  120-126 Months | -94.1 [-100.0 to -51.1]
  126-132 Months: number analyzed (Participants) | 6
  126-132 Months | -86.1 [-100.0 to -53.8]
  132-138 Months: number analyzed (Participants) | 2
  132-138 Months | -95.7 [-100.0 to -91.5]
Statistical Analysis 1: Comparison: Evaluation Group (Stimulation ON); Test type: Other; p < 0.05, Wilcoxon Signed Rank Test — For all 6-month periods, from 6 months through 9 years post-implant, p <0.05

3. Secondary Outcome: Responder Rate
Description: The proportion of subjects with greater than or equal to 50% reduction in total disabling seizures compared to pre-implant baseline.
Time Frame: 6 months post-implant through 9 years post-implant (8.5 years)
Population: N represents the number of subjects who have data during that period.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Evaluation Group (Stimulation ON)
Number analyzed (Participants) | 230
Percentage of patients
  6-12 Months: number analyzed (Participants) | 229
  6-12 Months | 33.2 [27.4 to 39.5]
  12-18 Months: number analyzed (Participants) | 229
  12-18 Months | 46.7 [40.4 to 53.2]
  18-24 Months: number analyzed (Participants) | 229
  18-24 Months | 47.6 [41.2 to 54.1]
  24-30 Months: number analyzed (Participants) | 223
  24-30 Months | 50.2 [43.7 to 56.7]
  30-36 Months: number analyzed (Participants) | 218
  30-36 Months | 56.4 [49.8 to 62.8]
  36-42 Months: number analyzed (Participants) | 218
  36-42 Months | 57.8 [51.2 to 64.2]
  42-48 Months: number analyzed (Participants) | 209
  42-48 Months | 61.2 [54.5 to 67.6]
  48-54 Months: number analyzed (Participants) | 201
  48-54 Months | 60.2 [53.3 to 66.7]
  54-60 Months: number analyzed (Participants) | 198
  54-60 Months | 61.1 [54.2 to 67.6]
  60-66 Months: number analyzed (Participants) | 190
  60-66 Months | 58.4 [51.3 to 65.2]
  66-72 Months: number analyzed (Participants) | 185
  66-72 Months | 67.0 [60.0 to 73.4]
  72-78 Months: number analyzed (Participants) | 181
  72-78 Months | 66.9 [59.7 to 73.3]
  78-84 Months: number analyzed (Participants) | 178
  78-84 Months | 65.7 [58.5 to 72.3]
  84-90 Months: number analyzed (Participants) | 171
  84-90 Months | 64.9 [57.5 to 71.7]
  90-96 Months: number analyzed (Participants) | 171
  90-96 Months | 70.2 [62.9 to 76.5]
  96-102 Months: number analyzed (Participants) | 168
  96-102 Months | 68.5 [61.1 to 75.0]
  102-108 Months: number analyzed (Participants) | 158
  102-108 Months | 70.9 [63.4 to 77.4]
  108-114 Months: number analyzed (Participants) | 110
  108-114 Months | 74.5 [65.7 to 81.8]
  114-120 Months: number analyzed (Participants) | 30
  114-120 Months | 66.7 [48.8 to 80.8]
  120-126 Months: number analyzed (Participants) | 12
  120-126 Months | 75.0 [46.8 to 91.1]
  126-132 Months: number analyzed (Participants) | 6
  126-132 Months | 83.3 [43.6 to 97.0]
  132-138 Months: number analyzed (Participants) | 2
  132-138 Months | 100.0 [34.2 to 100]

4. Secondary Outcome: QOLIE (Quality of Life in Epilepsy)
Description: QOLIE 89 (for English-speaking subjects) or QOLIE 31 P (for Spanish speaking subjects) scores collected at each year of follow-up after implantation of the RNS® System compared to the QOLIE 89 / QOLIE 31 P at pre-implant baseline. A QOLIE overall score was obtained using a weighted average of multi-item scale scores. The QOLIE overall score was converted to a T-score, a normally distributed scale with a mean score of 50 and standard deviation (SD) of 10. Higher scores reflect a better quality of life.
Time Frame: 1 year post-implant through 9 years post-implant (8 years)
Population: N represents the number of subjects who have data during that period.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Evaluation Group (Stimulation ON)
Number analyzed (Participants) | 230
Score on a scale
  Baseline: number analyzed (Participants) | 221
  Baseline | 46.1 (9.7)
  Year 1: number analyzed (Participants) | 216
  Year 1 | 49.2 (10.5)
  Year 2: number analyzed (Participants) | 208
  Year 2 | 49.3 (10.3)
  Year 3: number analyzed (Participants) | 208
  Year 3 | 48.8 (10.4)
  Year 4: number analyzed (Participants) | 194
  Year 4 | 48.1 (10.6)
  Year 5: number analyzed (Participants) | 186
  Year 5 | 48.4 (10.9)
  Year 6: number analyzed (Participants) | 165
  Year 6 | 48.4 (11.7)
  Year 7: number analyzed (Participants) | 165
  Year 7 | 47.4 (11.0)
  Year 8: number analyzed (Participants) | 156
  Year 8 | 47.9 (11.3)
  Year 9: number analyzed (Participants) | 150
  Year 9 | 47.2 (11.6)
Statistical Analysis 1: Comparison: Evaluation Group (Stimulation ON); Test type: Other; p < 0.0001, Generalized estimating equation (GEE); GEE estimated intercept = 48.0, 95% CI 2-sided [46.8 to 49.2]
Statistical Analysis 2: Comparison: Evaluation Group (Stimulation ON); Test type: Other; p = 0.6729, Generalized estimating equation (GEE); Slope = -0.0, 95% CI 2-sided [-0.2 to 0.1]

5. Secondary Outcome: Adverse Event Rate
Description: The rate of occurrence of any adverse event (AE) observed during the Long-term Treatment Investigation.
Time Frame: 6 months post-implant through 9 years post-implant (8.5 years)
Population: N represents the number of subjects who have data during that period.
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation Group (Stimulation ON)
Number analyzed (Participants) | 230
Participants | 228

ADVERSE EVENTS:
Time Frame: 6 months post-implant through 9 years post-implant (8.5 years)
Arm/Group | Evaluation Group (Stimulation ON)
All-Cause Mortality (participants affected / at risk) | 9/230
Serious Adverse Events (participants affected / at risk) | 177/230
Other Adverse Events (participants affected / at risk) | 228/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evaluation Group (Stimulation ON) (N=230)
EEG monitoring (Investigations) | 44 (63)
Implant site infection (Infections and infestations) | 26 (29)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 19 (22)
Tonic-clonic seizures increased (Nervous system disorders) | 12 (14)
Brain lobectomy (Surgical and medical procedures) | 11 (12)
Complex partial seizures increased (Nervous system disorders) | 10 (13)
Death (General disorders) | 9 (9)
Medical device removal (Surgical and medical procedures) | 9 (9)
Pneumonia (Nervous system disorders) | 9 (9)
Convulsive status epilepticus (Nervous system disorders) | 8 (10)
Implant site erosion (Injury, poisoning and procedural complications) | 8 (10)
Hospitalisation (Surgical and medical procedures) | 7 (9)
Suicide attempt (Psychiatric disorders) | 6 (7)
Depression suicidal (Psychiatric disorders) | 6 (6)
Postictal state (Nervous system disorders) | 6 (6)
Adverse drug reaction (General disorders) | 5 (5)
Psychotic disorder (Psychiatric disorders) | 5 (5)
Device lead damage (Injury, poisoning and procedural complications) | 5 (5)
Medical observation (Investigations) | 5 (6)
Nonconvulsive status epilepticus (Nervous system disorders) | 5 (9)
Nephrolithiasis (Renal and urinary disorders) | 5 (7)
Tonic-clonic seizures exacerbated (Nervous system disorders) | 5 (5)
Live birth (Product Issues) | 4 (4)
Hernia (General disorders) | 4 (4)
Complex partial seizures exacerbated (Nervous system disorders) | 4 (4)
Cerebral haemorrhage (Nervous system disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Angiogram cerebral (Investigations) | 4 (5)
Device lead revision (Injury, poisoning and procedural complications) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Lumbar vertebral fracture (dts) (Injury, poisoning and procedural complications) | 3 (3)
Investigation (Investigations) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Skin laceration (dts) (Injury, poisoning and procedural complications) | 3 (6)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (4)
Ovarian cyst (Reproductive system and breast disorders) | 3 (4)
Migraine (Nervous system disorders) | 3 (3)
Cranioplasty (Surgical and medical procedures) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Acute psychosis (Psychiatric disorders) | 2 (2)
Adenomyosis (Reproductive system and breast disorders) | 2 (2)
Appendicitis (Nervous system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cosmetic surgery (Surgical and medical procedures) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Head injury (dts) (Injury, poisoning and procedural complications) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Hip fracture (dts) (Injury, poisoning and procedural complications) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Intracranial hypotension (Injury, poisoning and procedural complications) | 2 (2)
Jaw fracture (dts) (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Postictal paralysis (Nervous system disorders) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (dts) (Injury, poisoning and procedural complications) | 2 (2)
Status epilepticus (Nervous system disorders) | 2 (2)
Subdural haematoma (dts) (Injury, poisoning and procedural complications) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Thermal burn (dts) (Injury, poisoning and procedural complications) | 2 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Traumatic intracranial haemorrhage (dts) (Injury, poisoning and procedural complications) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Implant site infection (dts) (Infections and infestations) | 2 (2)
Tracheostomy (Surgical and medical procedures) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vasectomy reversal (Surgical and medical procedures) | 1 (1)
Victim of crime (Social circumstances) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wrist fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Premature battery depletion (GB-2570) (Injury, poisoning and procedural complications) | 1 (1)
Premature battery depletion (RE-CR2450N) (Injury, poisoning and procedural complications) | 1 (1)
Device protrusion (Injury, poisoning and procedural complications) | 1 (1)
Device electrical finding (Injury, poisoning and procedural complications) | 1 (1)
Implant site discharge (General disorders) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Stitch abscess (Nervous system disorders) | 1 (1)
Simple partial seizures increased (sensory) (Nervous system disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intraventricular haemorrhage (dts) (Nervous system disorders) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Lumbar puncture (Investigations) | 1 (1)
Medical device implantation (LR) (Surgical and medical procedures) | 1 (1)
Medical device removal (LR) (Surgical and medical procedures) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Menicus lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Metastatic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuromyelitis optica (Nervous system disorders) | 1 (1)
Neutropenic infection (Infections and infestations) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Pelvic congestion (Reproductive system and breast disorders) | 1 (1)
Pelvic fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Pilonidal cyst (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyelonephritis (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Renal cell carcinoma state unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sepsis (Nervous system disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Simple partial seizures increased (motor) (Nervous system disorders) | 1 (1)
Skeletal injury (dts) (Injury, poisoning and procedural complications) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 1 (1)
Somatic delusion (Psychiatric disorders) | 1 (1)
Spinal fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Subarachnoid haemorrhage (dts) (Vascular disorders) | 1 (1)
Submandibular mass (General disorders) | 1 (1)
Suicidal behavior (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tonic-clonic seizures (Nervous system disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tracheal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Acute myeloid leukaemia (Blood and lymphatic system disorders) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Ankle fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Anticonvulsant drug level below therapeutic (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Arrhthmia supraventricular (Cardiac disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Aspiration (dts) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac syncope (Cardiac disorders) | 1 (1)
Cervical cyst (Reproductive system and breast disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Clostridium difficile colitis (Gastrointestinal disorders) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1)
Confusional state (Nervous system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (dts) (Injury, poisoning and procedural complications) | 1 (1)
Conversion disorders (Psychiatric disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drug dependence (Psychiatric disorders) | 1 (1)
Drug withdrawal headache (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1)
Epileptic psychosis (Psychiatric disorders) | 1 (1)
Face injury (dts) (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fall (dts) (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1)
Fractured skull depressed (Injury, poisoning and procedural complications) | 1 (1)
Gastrinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hand fracture (dts) (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoglycaemic coma (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evaluation Group (Stimulation ON) (N=230)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 115 (226)
Adverse drug reaction (General disorders) | 71 (113)
Implant site pain (General disorders) | 69 (103)
EEG monitoring (Investigations) | 44 (64)
Nasopharyngitis (Infections and infestations) | 42 (63)
Skin laceration (dts) (Injury, poisoning and procedural complications) | 41 (81)
Headache (Nervous system disorders) | 40 (51)
Influenza (Infections and infestations) | 33 (40)
Contusion (dts) (Injury, poisoning and procedural complications) | 31 (65)
Upper respiratory tract infection (Infections and infestations) | 30 (40)
Implant site infection (Infections and infestations) | 29 (34)
Urinary tract infection (Infections and infestations) | 29 (42)
Depression (Psychiatric disorders) | 28 (30)
Complex partial seizures increased (Nervous system disorders) | 25 (40)
Sinusitis (Nervous system disorders) | 25 (30)
Procedural pain (General disorders) | 24 (27)
Joint injury (Injury, poisoning and procedural complications) | 22 (26)
Rash (Skin and subcutaneous tissue disorders) | 22 (29)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Tonic-clonic seizures increased (Nervous system disorders) | 20 (25)
Diarrhoea (Gastrointestinal disorders) | 18 (19)
Vomiting (Gastrointestinal disorders) | 18 (20)
Vitamin D abnormal (Investigations) | 18 (18)
Joint injury (dts) (Injury, poisoning and procedural complications) | 18 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (19)
Tonic-clonic seizures exacerbated (Nervous system disorders) | 17 (19)
Head injury (dts) (Injury, poisoning and procedural complications) | 17 (25)
Complex partial seizures exacerbated (Nervous system disorders) | 16 (20)
Procedural headache (Injury, poisoning and procedural complications) | 16 (16)
Multiple injuries (dts) (Injury, poisoning and procedural complications) | 16 (38)
Insomnia (Nervous system disorders) | 16 (18)
Simple partial seizures (motor) (Nervous system disorders) | 15 (22)
Postictal state (Nervous system disorders) | 15 (15)
Drug hypersensitivity (Immune system disorders) | 14 (18)
Seasonal allergy (Immune system disorders) | 14 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (14)
Hypertension (Vascular disorders) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 13 (14)
Anxiety (Psychiatric disorders) | 13 (13)
Complex partial seizures (Nervous system disorders) | 13 (22)
Contusion (Injury, poisoning and procedural complications) | 13 (14)
Skin laceration (Injury, poisoning and procedural complications) | 13 (14)
Gastroenteritis (Nervous system disorders) | 13 (14)
Head injury (Injury, poisoning and procedural complications) | 13 (16)
Pneumonia (Infections and infestations) | 13 (16)
Road traffic accident (Injury, poisoning and procedural complications) | 13 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13)
Paraesthesia (Nervous system disorders) | 12 (12)
Nephrolithiasis (Renal and urinary disorders) | 12 (17)
Brain lobectomy (Surgical and medical procedures) | 11 (12)
Dizziness (Nervous system disorders) | 11 (12)
Ear infection (Infections and infestations) | 11 (14)
Temor (Nervous system disorders) | 11 (12)
Photopsia (Nervous system disorders) | 11 (15)
Simple partial seizures (sensory) (Nervous system disorders) | 11 (14)
Memory impairment (Nervous system disorders) | 11 (12)
Constipation (Gastrointestinal disorders) | 10 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (13)
Excoriation (dts) (Injury, poisoning and procedural complications) | 10 (35)
Dysaesthesia (Nervous system disorders) | 10 (11)
Agitation (Psychiatric disorders) | 9 (9)
Death (General disorders) | 9 (9)
Fall (dts) (Injury, poisoning and procedural complications) | 9 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 (9)
Tooth infection (Infections and infestations) | 9 (9)
Medical device removal (Surgical and medical procedures) | 9 (9)
Migraine (Nervous system disorders) | 9 (10)
Thermal burn (dts) (Injury, poisoning and procedural complications) | 9 (10)
Limb injury (Injury, poisoning and procedural complications) | 9 (9)
Convulsive status epilepticus (Nervous system disorders) | 8 (10)
Hypoaesthesia (Nervous system disorders) | 8 (10)
Implant site erosion (Injury, poisoning and procedural complications) | 8 (10)
Limb injury (dts) (Injury, poisoning and procedural complications) | 8 (9)
Toothache (Gastrointestinal disorders) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Pharyngitis (Infections and infestations) | 8 (9)
Simple partial seizures increased (sensory) (Nervous system disorders) | 8 (10)
Non-cardiac chest pain (General disorders) | 8 (9)
Depression suicidal (Psychiatric disorders) | 7 (7)
Device interaction (General disorders) | 7 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Hospitalisation (Surgical and medical procedures) | 7 (9)
Tooth extraction (Surgical and medical procedures) | 7 (7)
Nonconvulsive status epilepticus (Nervous system disorders) | 7 (11)
Psychotic disorder (Psychiatric disorders) | 7 (7)
Syncope (Nervous system disorders) | 7 (7)
Hypersensitivity (Immune system disorders) | 7 (9)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Vision blurred (Eye disorders) | 6 (6)
Clavicle fracture (dts) (Injury, poisoning and procedural complications) | 6 (8)
Conversion disorders (Psychiatric disorders) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Fatigue (General disorders) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 6 (6)
Hernia (General disorders) | 6 (6)
Muscle strain (Injury, poisoning and procedural complications) | 6 (6)
Oedema peripheral (General disorders) | 6 (6)
Procedural nausea (Injury, poisoning and procedural complications) | 6 (8)
Road traffic accident (dts) (Injury, poisoning and procedural complications) | 6 (6)
Simple partial seizures increased (motor) (Nervous system disorders) | 6 (9)
Sleep apnea (Nervous system disorders) | 6 (6)
Suicide attempt (Psychiatric disorders) | 6 (8)
Chest pain (General disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each Investigator and Institution agree that the 1st publication of study results shall be a joint, multi-center publication. Each Investigator, Coordinator, and Institution agree to submit publications to the RNS® System Study Publication Committee for review prior to submission for publication (at least 30 days for manuscripts and at least 7 days for abstracts) to assure that publication does not compromise the scientific integrity of the study or contain confidential NeuroPace information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT00572195/Prot_SAP_000.pdf